CLINICAL TRIAL: NCT05503615
Title: Investigation of the Effect of Instrument-Assisted Soft Tissue Mobilization Technique on Flexibility and Thickness in Gastrokinemius Muscle and Achilles Tendon With Compression Elastography Method in Healthy Individuals.
Brief Title: Investigation of the Effect of Instrument-Assisted Soft Tissue Mobilization Technique on Flexibility and Thickness by Compression Elastography Method in Healthy Individuals.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Muhammed Usame TAS, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ÜSAME TAŞ-003
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Instrument-assisted Soft Tissue Mobilization; Flexibility; Thickness; Compression Elastography; Rehabilitation
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Which leg of the individuals will be applied will be determined by the coin toss. After the money shot, the right leg will be applied when the writing comes, and the left leg will be applied when the tour comes. The leg to be applied includes the treatment group of the individuals; the other leg (the leg without application) will form the control group of individuals.
  Interventions: Other: Observational
- IASTM Treatment Group (Experimental): Which leg of the individuals will be applied will be determined by the coin toss. After the money shot, the right leg will be applied when the writing comes, and the left leg will be applied when the tour comes. The leg to be applied includes the treatment group of the individuals; the other leg (the leg without application) will form the control group of individuals.
  Interventions: Other: IASTM Technique Application

INTERVENTIONS:
Other: Observational — No application will be made to the control group.
  Arms: Control Group
Other: IASTM Technique Application — Instrument-assisted soft tissue mobilization will be applied to the legs of the individuals to be treated with ultrasound gel for 2 minutes.
  Arms: IASTM Treatment Group

SUMMARY:
Instrument-assisted soft tissue mobilization is an instrument-assisted soft tissue mobilization technique. It consists of stainless steel instrument designed to adapt to various tissues/shapes/curves of the body. The instruments were developed as an alternative to transverse friction massage. Stainless steel acts a bit like a diaposon when it comes into contact with fibrotic tissue. A resonance or reverberation in the instrument is created upon contact and transmitted through the instrument to the hands of the clinician. The application of heavy pressure (compared to light or medium pressure) using instruments has been proven to promote a greater fibroblastic response.

Instrument-assisted soft tissue mobilization is not used without insulation. It is imperative to use movement and strengthening in combination with soft tissue mobilization to promote tissue adaptation and remodeling. Mechanical loading has been shown to affect chondrocyte alignment and fibroblast activity with increased proteoglycan and collagen synthesis.

Elastography is an imaging method that allows the qualitative and quantitative evaluation of the biomechanical properties of tissues through USG. This imaging method provides information about the stiffness of the tissues independently of the acoustic impedance provided by B-mode examination and the vascular flow information provided by Doppler examination.

Compression elastography technique is based on the formation of strain (strain, displacement) in the compressed tissue. In hard tissues, displacement (strain) is less, while in soft tissues it is more. The displacement rates of the tissues are calculated by comparing the echo data obtained before and after the compression application. In compression elastography systems, the amount of pressure applied is indicated by an indicator on the screen.

The aim of this study was to investigate the effect of instrument-assisted soft tissue mobilization technique by compression elastography method on flexibility and thickness in gastrocnemius muscle and Achilles tendon in healthy individuals.

DETAILED DESCRIPTION:
In the study, iASTM will be applied to healthy individuals and the effect of this technique will be examined. Demographic information of individuals will be recorded and individuals will be evaluated in detail in terms of muscle and tendon flexibility and thickness.

The work plan; pre-treatment evaluation, followed by treatment and second evaluation immediately after the end of treatment. The data collection period is planned as 1,5 year.

ELIGIBILITY:
Inclusion Criteria:

1. Consists of healthy individuals between the ages of 18-35,
2. No history of orthopedic injury (muscle, tendon, joint capsule, ligament damage or peripheral neuropathy) in the lower extremities in the last 1 year,
3. Being able to express himself without cognitive, cognitive and mental problems,
4. Voluntarily agree to participate in the study.

Exclusion Criteria:

1. Injury to any lower extremity between measurements during the treatment process,
2. Having a BMI over 25,
3. Surgery or arthritis in the last 1 year,
4. Not being able or unwilling to do the tests,
5. Not wanting to leave of their own accord.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Muscle and Tendon Flexibility | Pre-treatment assessment.
  Compression elastography method will be used to measure flexibility in the gastrocnemius muscle and achilles tendon of individuals.
Evaluation of Muscle and Tendon Flexibility | Second assessment immediately after the end of the 10-minute treatment.
  Compression elastography method will be used to measure flexibility in the gastrocnemius muscle and achilles tendon of individuals.
Evaluation of Muscle and Tendon Thickness | Pre-treatment assessment.
  Compression elastography method will be used to measure thickness in the gastrocnemius muscle and achilles tendon of individuals.
Evaluation of Muscle and Tendon Thickness | Second assessment immediately after the end of the 10-minute treatment.
  Compression elastography method will be used to measure thickness in the gastrocnemius muscle and achilles tendon of individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Üsame TAŞ, Lecturer, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No